CLINICAL TRIAL: NCT05002244
Title: A Two-arm, Open-label, Single-sequence, Multiple-dose, Cross-over Phase 1 Study to Evaluate the Pharmacokinetic Interaction and Safety of CTL0801 and CTL0802 Compared to Coadministration in Healthy Adult Volunteers.
Brief Title: A Drug-Drug Interaction Study of CTL0801 and CTL0802 Compared to Coadministration in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L08-101
Record Dates: First submitted 2021-07-30; First posted 2021-08-12 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Health, Subjective
MeSH Terms: interventions — azilsartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): CTL0801 (Azilsartan) QD, 4days → CTL0801 (Azilsartan) + CTL0802 (Rosuvasatin) QD, 7days
  Interventions: Drug: CTL0801 (Azilsartan); Drug: CTL0801 (Azilsartan) + CTL0802 (Rosuvastatin)
- Arm B (Experimental): CTL0802 (Rosuvasatin) QD, 7days → CTL0801 (Azilsartan) + CTL0802 (Rosuvasatin) QD, 7days
  Interventions: Drug: CTL0802 (Rosuvastatin); Drug: CTL0801 (Azilsartan) + CTL0802 (Rosuvastatin)

INTERVENTIONS:
Drug: CTL0801 (Azilsartan) — CTL0801 (Azilsartan), single dose, daily, repeated oral administration
  Arms: Arm A
Drug: CTL0802 (Rosuvastatin) — CTL0802 (Rosuvastatin), single dose, daily, repeated oral administration
  Arms: Arm B
Drug: CTL0801 (Azilsartan) + CTL0802 (Rosuvastatin) — CTL0801 (Azilsartan) + CTL0802 (Rosuvastatin), single dose, daily, repeated oral administration

SUMMARY:
This is a two-arm, open-label, single-sequence, multiple-dose, cross-over phase 1 study to evaluate the interaction between two investigational drugs by comparing and analyzing the pharmacokinetic interaction and safety of CTL0801 and CTL0802 at steady state when administered alone or in combination with repeated oral doses in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A subject who weighs 50 kg or more (45 kg or more for women)
* A subject who does not have clinically significant congenital or chronic diseases
* A subject who is judged to be eligible to participate by the results of diagnostic tests by the principal investigator
* A subject and their partner who agree to use a medically appropriate method of contraception to exclude potential of pregnancy and not to provide sperm or ova from the first dose to 7 days after the last dose of the investigational drug
* A subject who voluntarily signs the consent form after hearing and understanding the purpose and content of this study, the characteristics of the investigational drugs, and expected adverse reactions

Exclusion Criteria:

* A subject who has a known digestive system, cardiovascular system, endocrine system, respiratory system, blood·tumor, infectious disease, kidney and genitourinary system, mental·nervous system, musculoskeletal system, immune system, otolaryngology, skin system, ophthalmic system or has any past history of them
* A subject who has a history of gastrointestinal surgery that may affect drug absorption (except simple appendectomy or hernia surgery) or has gastrointestinal diseases
* A subject who has taken drugs that induce or inhibit drug metabolizing enzymes such as barbiturates within 1 month of the first administration or has taken drugs that may affect the study within 10 days of the first administration (however, participation can be possible considering pharmacokinetic·pharmacodynamic characteristics such as interaction with concomitant drugs and half-life of concomitant drugs etc)
* A subject who has participated and administered other investigational drugs in other clinical trials or bioequivalence studies within 6 months of the first administration
* A subject who is judged ineligible for participation in this study by the principal investigator
* A female volunteer who is pregnant or lactating

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss | predose(0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and, 24 hours postdose
Cmax,ss | predose(0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and, 24 hours postdose

SECONDARY OUTCOMES:
Tmax,ss | predose(0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and, 24 hours postdose
Cmin,ss | predose(0 hour), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and, 24 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea